CLINICAL TRIAL: NCT00763789
Title: Local Anaesthesia and Remifentanil Sedation Versus Total Intravenous Anaesthesia for Hysteroscopic Surgery in an Ambulatory Surgery Department. A Randomized Clinical Trial.
Brief Title: Local Anaesthesia and Remifentanil Sedation Versus Total Intravenous Anaesthesia for Hysteroscopic Surgery in an Ambulatory Surgery Department.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Copenhagen University Hospital at Herlev (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H-D-2008-031
Record Dates: First submitted 2008-09-30; First posted 2008-10-01 (Estimated); Last update posted 2010-01-06 (Estimated); Status verified 2010-01

CONDITIONS: Conscious Sedation; Remifentanil; Hysteroscopic Surgery; Anesthesia Recovery Period; Ambulatory Surgery
Keywords: conscious sedation; remifentanil; hysteroscopic surgery; anesthesia recovery period; ambulatory surgery; patient satisfaction; length of stay
MeSH Terms: conditions — Patient Satisfaction | interventions — Anesthesia, Local

ARMS (2):
- 1 (Experimental): Local anaesthesia and remifentanil sedation
  Interventions: Other: local anaesthesia and remifentanil sedation
- 2 (Other): Total intravenous anaesthesia
  Interventions: Other: total intravenous anaesthesia

INTERVENTIONS:
Other: local anaesthesia and remifentanil sedation
  Arms: 1
Other: total intravenous anaesthesia
  Arms: 2

SUMMARY:
The purpose of this study is to compare a new method: the combination of conscious sedation with remifentanil (a shortlasting opioid drug) and local anaesthesia, with the traditional general anaesthesia for hysteroscopic surgery. The primary outcomes are: the time spent in the operation room, the time to full mobilisation postoperatively and the time to complete recovery postoperatively and the time to discharge. Secondary outcome: patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years,
* ASA classification I-II
* Speaks and writes danish
* Signed informed consent

Exclusion Criteria:

* ASA classification III-VI
* Emotional disorder - medically treated within a week before surgery
* Patients in risk of perioperative aspiration - who must be intubated
* BMI > 35
* Patients who have been using pain medicine within a week before surgery (except PCM and NSAID)
* Patients who have been using sleeping medicine or sedatives within a week before surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2008-08; Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
the total time spent in the operating room

CONTACTS AND LOCATIONS:
Locations (1):
- Copenhagen University Hospital Herlev, Copenhagen, Denmark